CLINICAL TRIAL: NCT04201730
Title: A Single Center, Open, Randomized Clinical Trial：Study on the Efficacy and Safety of Enhanced Recovery After Surgery （ERAS）in Gastrointestinal Cancer
Brief Title: Study on the Efficacy and Safety of Enhanced Recovery After Surgery （ERAS）in Gastrointestinal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jianbin Xiang, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2018-396
Record Dates: First submitted 2019-12-09; First posted 2019-12-17 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Enhanced Recovery After Surgery; Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ERAS (Experimental): Perioperative intervention with individual Enhanced Recovery After Surgery （ERAS）
  Interventions: Procedure: Enhanced Recovery After Surgery （ERAS）

INTERVENTIONS:
Procedure: Enhanced Recovery After Surgery （ERAS） — Preoperative education，Preoperative nutritional support，Preoperative bowel preparation，Preventative applying of antibiotics，Intraoperative warming，Goal-directed fluid therapy，Postoperative analgesia，Postoperative diet, drainage and activity management，Prevention of deep vein thrombosis.

SUMMARY:
At present, there are more and more reports about enhanced recovery after surgery（ERAS）in China, but there is no ERAS treatment standard for gastrointestinal cancer, and there are many factors limiting the development of ERAS. In recent years, due to the development of minimally invasive technology, the establishment of evidence-based medicine model and the development of MDT, it makes a good solid foundation for the clinical application of ERAS. The implementation of ERAS requires the cooperation of surgeons, anesthesia management, nursing, rehabilitation and other teams. As an individualized treatment mode, ERAS focuses on the optimization of treatment for different individuals in order to acquire the best benefit of patients. Therefore, the concept of ERAS is still in the process of continuous improvement and development in China, hoping to explore the Chinese ERAS clinical pathway for gastrointestinal cancer. The purpose of this study is to optimize the clinical pathway of ERAS in the perioperative period of gastrointestinal cancer, and to evaluate the effectiveness and safety of ERAS in gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent
* Preoperative pathology confirmed gastric cancer or colorectal cancer
* Age: 18-70 years, men or women
* According to NCCN guidelines, it is not Stage IV tumor
* Perform radical gastrectomy or radical colon cancer surgery (CME) or radical rectal cancer surgery (TME);
* ASA I-III
* Receive no radiotherapy or chemotherapy before operation
* The subjects can describe the symptoms objectively and keep the follow-up plan

Exclusion Criteria:

* Preoperative pathology confirmed no gastric cancer / no colorectal cancer (such as rectal neuroendocrine tumor, lymphoma, etc.)
* Stage IV or Radical resection can't be performed
* Emergency operation
* Can't cooperate with clinical data collection
* General condition is intolerable to operation
* Serious diseases, including heart function ≥ level II, respiratory function insufficiency, liver and kidney function insufficiency, and blood system diseases
* Patients participate in other clinical trials at the same time
* Pregnant or perinatal women
* Other malignant tumors
* History of mental illness
* Had a history of severe trauma within 4 weeks before admission
* Less than 6 months after other level 4 operations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Hospitalization Days | Postoperative up to 2 weeks
Time of getting out of bed after operation | Postoperative 7 days
The time to first flatus | Postoperative 7 days

SECONDARY OUTCOMES:
Expenses on medical treatment, medicine and hospitalization | On discharge, Postoperative up to 2 weeks
Incidence of postoperative complications | Postoperative 3 months、6 months、1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilmore DW, Kehlet H. Management of patients in fast track surgery. BMJ. 2001 Feb 24;322(7284):473-6. doi: 10.1136/bmj.322.7284.473. No abstract available. PMID 11222424
- [Result] Lee SM, Kang SB, Jang JH, Park JS, Hong S, Lee TG, Ahn S. Early rehabilitation versus conventional care after laparoscopic rectal surgery: a prospective, randomized, controlled trial. Surg Endosc. 2013 Oct;27(10):3902-9. doi: 10.1007/s00464-013-3006-4. Epub 2013 May 25. PMID 23708720
- [Result] Kehlet H. Fast-track surgery-an update on physiological care principles to enhance recovery. Langenbecks Arch Surg. 2011 Jun;396(5):585-90. doi: 10.1007/s00423-011-0790-y. Epub 2011 Apr 6. PMID 21468643
- [Result] Aarts MA, Okrainec A, Glicksman A, Pearsall E, Victor JC, McLeod RS. Adoption of enhanced recovery after surgery (ERAS) strategies for colorectal surgery at academic teaching hospitals and impact on total length of hospital stay. Surg Endosc. 2012 Feb;26(2):442-50. doi: 10.1007/s00464-011-1897-5. Epub 2011 Oct 20. PMID 22011937
- [Result] Jie B, Jiang ZM, Nolan MT, Zhu SN, Yu K, Kondrup J. Impact of preoperative nutritional support on clinical outcome in abdominal surgical patients at nutritional risk. Nutrition. 2012 Oct;28(10):1022-7. doi: 10.1016/j.nut.2012.01.017. Epub 2012 Jun 5. PMID 22673593
- [Result] Li P, Fang F, Cai JX, Tang D, Li QG, Wang DR. Fast-track rehabilitation vs conventional care in laparoscopic colorectal resection for colorectal malignancy: a meta-analysis. World J Gastroenterol. 2013 Dec 21;19(47):9119-26. doi: 10.3748/wjg.v19.i47.9119. PMID 24379639
- [Result] Li YJ, Huo TT, Xing J, An JZ, Han ZY, Liu XN, Zhao QC. Meta-analysis of efficacy and safety of fast-track surgery in gastrectomy for gastric cancer. World J Surg. 2014 Dec;38(12):3142-51. doi: 10.1007/s00268-014-2690-0. PMID 25228170
- [Result] Spanjersberg WR, van Sambeeck JD, Bremers A, Rosman C, van Laarhoven CJ. Systematic review and meta-analysis for laparoscopic versus open colon surgery with or without an ERAS programme. Surg Endosc. 2015 Dec;29(12):3443-53. doi: 10.1007/s00464-015-4148-3. Epub 2015 Mar 24. PMID 25801106
- [Result] Ni TG, Yang HT, Zhang H, Meng HP, Li B. Enhanced recovery after surgery programs in patients undergoing hepatectomy: A meta-analysis. World J Gastroenterol. 2015 Aug 14;21(30):9209-16. doi: 10.3748/wjg.v21.i30.9209. PMID 26290648
- [Result] Sammour T, Zargar-Shoshtari K, Bhat A, Kahokehr A, Hill AG. A programme of Enhanced Recovery After Surgery (ERAS) is a cost-effective intervention in elective colonic surgery. N Z Med J. 2010 Jul 30;123(1319):61-70. PMID 20717178